CLINICAL TRIAL: NCT02156128
Title: Study of Subjective Memory Complaints, Objective Memory Performance and Cognitive Training in Patients With Complex Symptom Disorders
Brief Title: Subjective Memory Complaints, Objective Memory Performance and Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100878
Record Dates: First submitted 2014-06-03; First posted 2014-06-05 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Fatigue Syndrome, Chronic; Chronic Pain; Anxiety Disorders; Depressive Disorder; Sleep Disorders
Keywords: Cognitive therapy
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Chronic Pain; Anxiety Disorders; Depressive Disorder; Sleep Wake Disorders | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cogmed (Experimental): Participants in a 3,5 week vocational rehabilitation program (containing cognitive therapy and physical exercise) are instructed to use a computer-based working memory training program (named CogMed) each weekday (5 days a week) for 5 weeks. Each training session consists of 8 different tasks and lasts 40-50 minutes.
  Interventions: Behavioral: Cogmed working memory training
- Control group (Active Comparator): These subjects will participate in the vocational rehabilitation program for 3,5 weeks. The program includes cognitive therapy (ACT) and physical activity, but no working memory training.
  Interventions: Behavioral: Control group

INTERVENTIONS:
Behavioral: Cogmed working memory training
  Arms: Cogmed
Behavioral: Control group
  Arms: Control group

SUMMARY:
The aim of this study is to examine if repetitive computerized cognitive training improves working memory in patients who are on sick leave due to complex symptom disorders (chronic pain, chronic fatigue, anxiety, depression and or sleep disorders), and whether effects of cognitive control training transfer to other tasks.

ELIGIBILITY:
Inclusion Criteria:

* on sick leave due to complex symptom disorders: chronic pain, chronic fatigue, anxiety, depression and/or sleep disorders
* on sick leave for at least eight weeks.

Exclusion Criteria:

* severe mental disorder
* acute psychosis
* ongoing manic episode
* suicidal ideation
* ongoing abuse of alcohol or any other substance.
* not able to communicate in Norwegian

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2013-10; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Working memory capacity | 7 weeks
  Objective memory performance as assessed by a sample of neuropsychological tests from Cambridge Cognition - Cantab tests (Spatial Working Memory (SWM), One Touch Stockings of Cambridge (OTS), Stop Signal Task (SST)) Including Paced Auditory Serial Addition Test (PASAT).

SECONDARY OUTCOMES:
Subjective memory complaints (SMC) | 7 weeks
  Subjective memory complaints (SMC) are measured by a self-report questionnaire "The Everyday Memory Questionnaire" We estimate prevalence of subjective memory complaints and examine the correspondence between SMC and symptoms of depression, anxiety, sleep disturbances, chronic fatigue and chronic pain.
Transfer to inhibition | 7 weeks
  Transfer to inhibition is demonstrated by significantly reduced Stop Signal Reaction Time on The Stop Signal Task

CONTACTS AND LOCATIONS:
Overall Officials: Nils I Landrø, Prof, Study Director — Norwegian University of Science and Technology
Locations (1):
- NKSS Nasjonal kompetansetjeneste for sammensatte symptomlidelser, Trondheim, Norway

REFERENCES:
- [Result] Aasvik JK, Woodhouse A, Stiles TC, Jacobsen HB, Landmark T, Glette M, Borchgrevink PC, Landro NI. Effectiveness of Working Memory Training among Subjects Currently on Sick Leave Due to Complex Symptoms. Front Psychol. 2017 Jan 6;7:2003. doi: 10.3389/fpsyg.2016.02003. eCollection 2016. PMID 28111555